CLINICAL TRIAL: NCT03473366
Title: Safety and Efficacy of the Tao Facemask for Positive Pressure Ventilation in the Patients With Significantly Elevated BMIs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Carey Brewbaker, Assistant Professor Anesthesiology, Medical University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pro00073465
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Anesthesia Induction Ventilation

STUDY DESIGN:
Intervention Model Description: The sequence of standard vs Tao mask will be determined by random number generator. Mask ventilation will be scored with both masks before and after the standard administration of paralytic medication. The duration of the study procedures is variable but would last approximately 30-60 seconds, seldom exceeding 5 minutes additional time to the study patient from what is necessary in a non-study patient. The number of ventilations to achieve adequate ventilation is variable with both the standard mask and the Tao mask. After grading mask ventilation the study intervention is complete and the remainder of surgical and anesthesia care will be based on the clinical needs and decisions of the care team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tao Mask (Experimental): All anesthesiologists and CRNAs will view an instructional video on the use of the Tao Mask. Following induction of general anesthesia with the standard of care sequence of medications, each patient will then have mask ventilation performed and graded (Han and Warters Scales).Mask ventilation will be scored before and after the standard administration of paralytic medication.
  Interventions: Device: Tao Mask
- Standard Mask (Active Comparator): Following induction of general anesthesia with the standard of care sequence of medications, each patient will then have mask ventilation performed and graded (Han and Warters Scales).Mask ventilation will be scored before and after the standard administration of paralytic medication.
  Interventions: Device: Standard Mask

INTERVENTIONS:
Device: Tao Mask — All anesthesiologists and CRNAs will view an instructional video on the use of the Tao Mask. Following induction of general anesthesia with the standard of care sequence of medications, each patient will then have mask ventilation performed and graded (Han and Warters Scales).
  Arms: Tao Mask
Device: Standard Mask — Following induction of general anesthesia with the standard of care sequence of medications, each patient will then have mask ventilation performed and graded (Han and Warters Scales).Mask ventilation will be scored before and after the standard administration of paralytic medication.
  Arms: Standard Mask

SUMMARY:
The Tao Mask is a new novel facemask for positive pressure ventilation which has recently been demonstrated (MUSC study Pro00047645) to have superior performance to our conventional (standard) positive pressure mask in a random distribution of patients with experiences users. This additional study will extend our investigation of the new masks capabilities by studying it's performance in the morbidly obese - which are more challenging patients to ventilate by mask. Our hypothesis is that the Tao mask will be even more effective in this challenging population than in the random distribution of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years.
2. BMI of >40.
3. Patients having elective surgery (designated by priority level of 5) requiring general endotracheal anesthesia.

Exclusion Criteria:

1. Need for awake intubation based on standard preoperative evaluation by the attending anesthesiologist.
2. Increased risk for aspiration of gastric contents due to full stomach, pregnancy, gastro-esophageal reflux disease, and/or hiatal hernia as identified during the pre-operative assessment.
3. Previous tracheostomy procedure.
4. Patient is cognitively incapable of providing their consent for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Tao Scale Score | one year
  The primary outcome will be the Tao Scale Score for each mask, compared between patients

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Brewbaker CL, Wilson PR, McSwain JR, Tobin CD, Bridges KH, Roberts LL, Wilson DA, Skorke CA, Brown TA. Safety and efficacy of the Tao facemask for positive pressure ventilation in morbidly obese patients. J Perioper Pract. 2025 Dec;35(12):615-624. doi: 10.1177/17504589241268247. Epub 2024 Sep 18. PMID 41263061